CLINICAL TRIAL: NCT04540991
Title: Genotoxicity Assessment of Dental Implants in Gingival Epithelial Cells
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daniel Jerković (Other)
Responsible Party: Sponsor-Investigator, Daniel Jerković, DMD, University of Zagreb
Organization: University of Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 003-08/20-03/0005
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Genotoxicity
Keywords: implantology; genotoxicity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankylos dental implant group (Active Comparator): Patients are divided into two groups depending on the dental implant system used in the therapy. Ankylos dental implants (Dentsplay Sirona, Charlotte, USA) areused in the first group of patients.
  Interventions: Procedure: implant placement; Procedure: gingiva former placement; Diagnostic Test: Collecting gingival epithelial cellsusing the swab technique
- Dentium SuperLine implant group (Active Comparator): Patients are divided into two groups depending on the dental implant system used in the therapy. Dentium SuperLine implants (Dentium Co., Seoul, Korea) is used in the second group of patients-.
  Interventions: Procedure: implant placement; Procedure: gingiva former placement; Diagnostic Test: Collecting gingival epithelial cellsusing the swab technique

INTERVENTIONS:
Procedure: implant placement — The implants are placed in accordance with each implant system manufacturer's instructions and the treatment were performed according to the patient's standards and indications. Surgical procedures on all patients are performed by the same operator with the same surgical approach, protocol and instrumentation.
Procedure: gingiva former placement — Gingiva former are placed in accordance with each implant system manufacturer's instructions and the treatment were performed according to the patient's standards and indications. Surgical procedures of oppeninf implant cower and gingiva former placement on all patients are performed by the same operator with the same surgical approach, protocol and instrumentation.
Diagnostic Test: Collecting gingival epithelial cellsusing the swab technique — Samples of gingival epithelial cells are collected from each participant's implementation site using the swab technique at three different time points: a control swab is taken just before the placement of the dental implant (T0); the second swab is taken 90 days after implantation meaning immediately before placement of the gingiva former (T1); and the third swab is taken 21 days after placement of the gingiva former (T2).

SUMMARY:
Due to the strong correlation between genotoxicity and carcinogenesis, it is necessary to clarify the potential genotoxic effects of titanium dental implant systems. As most dental materials release small amounts of several elements into the oral cavity, proper regulations have to guarantee that the concern from genotoxicity/mutagenicity of dental materials is annulated or at the lowest possible level. Thus, further biocompatibility records are needed in order to evaluate the comprehensive risks of these compounds. In a view of the above-mentioned data, the aim of this in vivo study is to evaluate genotoxic and cytotoxic potential of implants and gingiva formers from two different implant systems in gingival epithelial cells.

Exfoliated gingival cells will be taken from 80 participants before and after 90 days of dental implant insertion, and 21 days following gingiva former placement. DNA damage will be analyzed using the micronucleus test. Tested dental implants will be Ankylos and Dentium, with corresponding gingival former.

DETAILED DESCRIPTION:
Patients are divided into two groups depending on the dental implant system used in the therapy. Ankylos dental implants (Dentsplay Sirona, Charlotte, USA) are used in the first group of patients and Dentium SuperLine (Dentium Co., Seoul, Korea) in the second group.

The implants are placed in accordance with each implant system manufacturer's instructions and the treatment were performed according to the patient's standards and indications. Surgical procedures on all patients are performed by the same operator with the same surgical approach, protocol and instrumentation.

The surgeries are performed under local anesthesia and systemic antibiotics were given according to standard procedure. To ensure post-surgical oral hygiene, patients are advised to rinse the oral cavity with chlorhexidine until the day of sutures' removal. The sutures are removed10 day after implantation. The implants are healing by being submerged for 12 weeks based on the surgeon's clinical judgment, indications given and the need and preference of the patients. After healing, gingiva formers are placed.

Sample collection and a micronucleus assay in gingival epithelial cells To reduce individual variations, patients are observed longitudinally and each subject is served as their own control. Samples of gingival epithelial cells are collected from each participant's implementation site using the swab technique at three different time points: a control swab is taken just before the placement of the dental implant (T0); the second swab is taken 90 days after implantation meaning immediately before placement of the gingiva former (T1); and the third swab is taken 21 days after placement of the gingiva former (T2).

One hour before the sampling, the participants abstain from consuming any food and drinks. After rinsing of the oral cavity 3 times with tepid water to remove exfoliated cells, a T0 swab is taken by gently brushing the gingiva around place indicated for implant placement and later T1 and T2 around implant with a cytobrush (Cytobrush Plus; GmbH. Dietramszell-Linden, Germany). The samples are subsequently applied to coded laboratory glass slides.

The cells applied to microscopic slides are allowed to air-dry and fixed in methanol (80% v/v) at 4°C for 20 minutes. Staining is conducted with 5% Giemsa solution for 10 minutes. Afterward, the slides are rinsed with aqua distillate and air dry. The slides are examined under Olympus CX40 light microscope (Olympus. Tokyo. Japan) with 400× magnification, and each micronucleus and other nuclear anomalies are additionally verified under 1000× magnification. Two replicate slides are prepared for each subject and 1000 epithelium cells per preparation were analyzed for each sampling time.

Nuclear anomalies, such as micronucleus, karyorrhexis (nuclear disintegration indicating apoptosis), karyolysis (dissolution of the nucleus mostly indicating necrosis and apoptosis), pyknosis (nuclear shrinkage due to apoptosis), condensed chromatin (DNA complexed with proteins and apoptosis), nuclear buds (precursors of micronuclei, or high density of DNA repair complexes) and broken eggs (nuclei that appear cinched, binucleated cells (indicating impaired velocity of cell proliferation)) are estimated and qualified.

ELIGIBILITY:
Inclusion Criteria:

* absence of a single tooth in the mandibular molar or premolar region
* belonging to ASA I or ASA II group
* absence of titanium hypersensitivity
* absence of prosthetic restoration/replacement or orthodontic appliances in the oral cavity, -absence of oral precancerous lesions
* no history of radiation in the head and neck area
* absence of bisphosphonates and corticosteroids used in therapy.

Exclusion Criteria:

* presence of systemic disease (e.g. uncontrolled diabetes, oral mucosal diseases, untreated gingivitis and periodontitis, endodontic lesions)
* pocket depths ≥ 4 mm on adjacent teeth
* bruxism
* poor oral hygiene
* pregnant and lactating women
* taking of antibiotics in the last three months
* taking any other pharmaceutics that have been proved to elevate DNA damage,
* underwent medical radiation diagnostics
* using mouthwash that contain alcohol
* history of radiation in the head and neck area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-03-20 (Estimated); Study Completion 2022-04-25 (Estimated)

PRIMARY OUTCOMES:
Cytotoxic and/or genotoxic | 1 year
  Evaluation of the cytotoxic and genotoxic alterations in gingival epithelial cells after application of titanium-based dental implant system

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jerkovic, DMD, Principal Investigator — University of Split, School of Medicine
Locations (1):
- School of Medicine, University of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piraccini BM, Urciuoli B, Starace M, Tosti A, Balestri R. Yellow nail syndrome: clinical experience in a series of 21 patients. J Dtsch Dermatol Ges. 2014 Feb;12(2):131-7. doi: 10.1111/ddg.12216. Epub 2013 Oct 18. PMID 24134631
- [Background] Berglund F, Carlmark B. Titanium, sinusitis, and the yellow nail syndrome. Biol Trace Elem Res. 2011 Oct;143(1):1-7. doi: 10.1007/s12011-010-8828-5. Epub 2010 Sep 1. PMID 20809268
- [Background] Sidambe AT. Biocompatibility of Advanced Manufactured Titanium Implants-A Review. Materials (Basel). 2014 Dec 19;7(12):8168-8188. doi: 10.3390/ma7128168. PMID 28788296
- [Background] Maloney WJ, Smith RL, Castro F, Schurman DJ. Fibroblast response to metallic debris in vitro. Enzyme induction cell proliferation, and toxicity. J Bone Joint Surg Am. 1993 Jun;75(6):835-44. doi: 10.2106/00004623-199306000-00005. PMID 8314824
- [Background] Wang JJ, Sanderson BJ, Wang H. Cyto- and genotoxicity of ultrafine TiO2 particles in cultured human lymphoblastoid cells. Mutat Res. 2007 Apr 2;628(2):99-106. doi: 10.1016/j.mrgentox.2006.12.003. Epub 2006 Dec 15. PMID 17223607
- [Background] Okuda-Shimazaki J, Takaku S, Kanehira K, Sonezaki S, Taniguchi A. Effects of titanium dioxide nanoparticle aggregate size on gene expression. Int J Mol Sci. 2010 Jun 7;11(6):2383-92. doi: 10.3390/ijms11062383. PMID 20640159
- [Background] Camacho-Alonso F, Sanchez-Siles M, Gilbel-del Aguila O. No Evidence of Genotoxic Damage in a Group of Patients with Titanium Dental Implants and Different Metal Restorations in the Oral Cavity. Clin Implant Dent Relat Res. 2015 Aug;17(4):811-21. doi: 10.1111/cid.12163. Epub 2013 Oct 17. PMID 24131612
- [Background] Karahalil B, Kadioglu E, Tuzuner-Oncul AM, Cimen E, Emerce E, Kisnisci RS. Micronucleus assay assessment of possible genotoxic effects in patients treated with titanium alloy endosseous implants or miniplates. Mutat Res Genet Toxicol Environ Mutagen. 2014 Jan 15;760:70-2. doi: 10.1016/j.mrgentox.2013.10.005. Epub 2013 Nov 1. PMID 24189049
- [Background] de Barros Lucena GA, de Molon RS, Moretti AJ, Shibli JA, Rego DM. Evaluation of Microbial Contamination in the Inner Surface of Titanium Implants Before Healing Abutment Connection: A Prospective Clinical Trial. Int J Oral Maxillofac Implants. 2018 Jul/Aug;33(4):853-862. doi: 10.11607/jomi.5817. PMID 30025002
- [Background] Makihira S, Mine Y, Nikawa H, Shuto T, Iwata S, Hosokawa R, Kamoi K, Okazaki S, Yamaguchi Y. Titanium ion induces necrosis and sensitivity to lipopolysaccharide in gingival epithelial-like cells. Toxicol In Vitro. 2010 Oct;24(7):1905-10. doi: 10.1016/j.tiv.2010.07.023. Epub 2010 Aug 1. PMID 20682337
- [Background] Harris BH, Kohles SS. Effects of mechanical and thermal fatigue on dental drill performance. Int J Oral Maxillofac Implants. 2001 Nov-Dec;16(6):819-26. PMID 11769832
- [Background] Souza JCM, Henriques M, Teughels W, Ponthiaux P, Celis JP, Rocha LA. Wear and corrosion interactions on titanium in oral environment: literature review. J Bio Tribo Corros. 2015;1:1-13.
- [Background] Broggini N, McManus LM, Hermann JS, Medina R, Schenk RK, Buser D, Cochran DL. Peri-implant inflammation defined by the implant-abutment interface. J Dent Res. 2006 May;85(5):473-8. doi: 10.1177/154405910608500515. PMID 16632764
- [Background] Superline | Products | Dentium [Internet]. Dentiumusa.com. 2020 [citirano 21.6.2020.]. Dostupno na: http://dentiumusa.com/products/dentalimplant/superline.htm
- [Background] Ankylos | Dentsply Sirona [Internet]. Dentsplysirona.com. 2020 [citirano 21.6.2020]. Dostupno na: https://www.dentsplysirona.com/enus/categories/implantology/ankylos.html
- [Background] Thomas P, Holland N, Bolognesi C, Kirsch-Volders M, Bonassi S, Zeiger E, Knasmueller S, Fenech M. Buccal micronucleus cytome assay. Nat Protoc. 2009;4(6):825-37. doi: 10.1038/nprot.2009.53. Epub 2009 May 7. PMID 19444240
- [Background] Holland N, Bolognesi C, Kirsch-Volders M, Bonassi S, Zeiger E, Knasmueller S, Fenech M. The micronucleus assay in human buccal cells as a tool for biomonitoring DNA damage: the HUMN project perspective on current status and knowledge gaps. Mutat Res. 2008 Jul-Aug;659(1-2):93-108. doi: 10.1016/j.mrrev.2008.03.007. Epub 2008 Apr 11. PMID 18514568
- [Background] Visalli G, Baluce B, La Maestra S, Micale RT, Cingano L, De Flora S, Di Pietro A. Genotoxic damage in the oral mucosal cells of subjects carrying restorative dental fillings. Arch Toxicol. 2013 Dec;87(12):2247-8. doi: 10.1007/s00204-013-1155-9. Epub 2013 Nov 16. No abstract available. PMID 24241249
- [Background] Thomas P, Bandl WD, Maier S, Summer B, Przybilla B. Hypersensitivity to titanium osteosynthesis with impaired fracture healing, eczema, and T-cell hyperresponsiveness in vitro: case report and review of the literature. Contact Dermatitis. 2006 Oct;55(4):199-202. doi: 10.1111/j.1600-0536.2006.00931.x. PMID 16958916
- [Background] Oshida Y, Tuna EB, Aktoren O, Gencay K. Dental implant systems. Int J Mol Sci. 2010 Apr 12;11(4):1580-678. doi: 10.3390/ijms11041580. PMID 20480036
- [Background] Branemark PI, Hansson BO, Adell R, Breine U, Lindstrom J, Hallen O, Ohman A. Osseointegrated implants in the treatment of the edentulous jaw. Experience from a 10-year period. Scand J Plast Reconstr Surg Suppl. 1977;16:1-132. No abstract available. PMID 356184
- [Background] Pjetursson BE, Zarauz C, Strasding M, Sailer I, Zwahlen M, Zembic A. A systematic review of the influence of the implant-abutment connection on the clinical outcomes of ceramic and metal implant abutments supporting fixed implant reconstructions. Clin Oral Implants Res. 2018 Oct;29 Suppl 18:160-183. doi: 10.1111/clr.13362. PMID 30306682